CLINICAL TRIAL: NCT00710372
Title: A Double Blind, Randomized, Placebo Controlled, Parallel Group, Dose-Titration Phase II Study to Evaluate Safety and Tolerability, Pharmacodynamic Effects and Efficacy of an Anti-Angiotensin II Vaccine (CYT006-AngQb) in Patients With Mild to Moderate Essential Hypertension
Brief Title: Safety, Tolerability and Efficacy of a Vaccine Against Essential Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cytos Biotechnology AG (Industry)
Responsible Party: Cytos Biotechnology, Cytos Biotechnology AG
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CYT006-AngQb 03; EudraCT No.: 2007-007516-28
Record Dates: First submitted 2008-07-03; First posted 2008-07-04 (Estimated); Last update posted 2010-11-15 (Estimated); Status verified 2010-11

CONDITIONS: Mild Essential Hypertension; Moderate Essential Hypertension
MeSH Terms: interventions — CYT006-AngQb

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): CYT006-AngQb
  Interventions: Biological: CYT006-AngQb
- 2 (Placebo Comparator)
  Interventions: Biological: CYT006-AngQb

INTERVENTIONS:
Biological: CYT006-AngQb — s.c. injection

SUMMARY:
The study medication CYT006-AngQb is a vaccine, consisting of angiotensin II (Ang II), the naturally occurring octapeptide coupled onto the surface of virus-like particles (VLP). This form of presenting Ang II to the immune system induces a B-cell mediated immune response characterized by the generation of specific antibodies (IgG and IgM) against Ang II. The CYT006-AngQb vaccine is administered by subcutaneous (s.c.) injection. Immunization against angiotensin II may offer a valuable alternative to conventional drugs for the treatment of hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild to moderate essential hypertension (Grade I and Grade II) with mean sitting office SBP =140-179 mmHg and/or mean sitting office DBP = 90 -109 mmHg on 2 consecutive visits (screening and V1).
* Daytime blood pressure above threshold for definition of hypertension in the baseline ABPM measurement (SBP >135 mmHg).
* Stable baseline blood pressure confirmed on 2 consecutive visits (screening and V1). (Changes <20mmHg for sitting office SBP and <10mmHg for mean sitting office DPB).
* Patients without current antihypertensive therapy. Patients on previous mono-antihypertensive therapy, who can safely stop their medication
* Patient is willing and able to comply with all trial requirements and procedures.

Exclusion Criteria:

* Patients with "very high added risk" according to 2007 Guidelines for the Management of Arterial Hypertension (Journal of Hypertension, 2007, 25:1105- 1187), i.e. those with:grade III hypertension (mean sitting office SBP

  * 180mmHg and/or meansitting DBP ≥110mmHg/history or presence of established cardiovascular or renal disease (Ischemic stroke, cerebral hemorrhage, transient ischemic attack)/ Myocardial infarction, angina pectoris, coronary re-vascularization/ clinically relevant heart failure (NYHA class II-IV)/ Peripheral artery disease/ Diabetic nephropathy
* Electrocardiographic confirmed left ventricular hypertrophy
* Increased plasma creatinine
* Diabetes mellitus type I, history, presence or new diagnosis of diabetes mellitus type II.
* Postural hypotension at screening
* Arrhythmias that would interfere with the oscilloscopic measurement of the blood pressure.
* Known autoimmune disease.
* Severe allergy.
* Pregnancy or breastfeeding.
* Women in childbearing age that are not surgically sterilized.
* Patients with a history or current positive test for HIV infection, AIDS, or other immunosuppressive disorders; hepatitis B or C.
* Current diagnosis or history of malignancy.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2008-06; Primary Completion 2009-07 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Adverse events: quality, quantity, severity | throughout complete study until week 48

SECONDARY OUTCOMES:
Change in daytime, nighttime and 24h ambulatory blood pressure from baseline | 24 hours
anti-Angio II IgG antibody titer | throughout complete study until week 48
Level of RAS Biomarkers (concentrations of plasma renin, angiotensinII and aldosterone) | 24 h

CONTACTS AND LOCATIONS:
Locations (1):
- Cytos Biotechnology (Sponsor's Headquarter), Schlieren, Switzerland